CLINICAL TRIAL: NCT02408640
Title: Internet-Based Treatment for Individuals With Regular Cannabis Use: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Kristina Sinadinovic, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/1374-31/5-1
Record Dates: First submitted 2015-03-26; First posted 2015-04-03 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Cannabis
Keywords: Internet-Based; Treatment
MeSH Terms: conditions — Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Intervention group (Experimental): Individuals randomized to the intervention group will directly after randomization answer questions about alcohol and drug use (other than alcohol and cannabis), depression, anxiety, a sense of context and whether they during the last 12 months has received professional help to reduce or quit their cannabis use or during the same period have raised this issue with their relatives or friends.
  Further, they will fill out a survey about Internet-based services for individuals who wish to reduce or quit their cannabis use. The study participants will then be informed that they, within two days, will gain access to an internet based treatment program designed to help them quit their cannabis use and that they through the program will be able to communicate with a therapist. Within the next two days, they will gain access to the internet-based treatment program, they will have access to it for two months and they will be contacted again after three months to complete the follow-up.
  Interventions: Behavioral: Cannabishjalpen.se
- Control group (No Intervention): Individuals randomized to the control group will undergo exactly the same procedure as the intervention group. The difference is that the control group will be informed that they in about three months will gain access to an internet based treatment program designed to help them quit their cannabis use (i.e. when the data collection for follow-up is completed).
  Otherwise, participants in both groups will have the opportunity to use factual information that is available to everyone on Cannabishjalpen.se.

INTERVENTIONS:
Behavioral: Cannabishjalpen.se
  Arms: Intervention group

SUMMARY:
The aim of this randomized controlled trial is to investigate the effects of a Swedish Internet-based treatment program for individuals from the general population with a regular cannabis use.

The primary hypothesis to be tested is that the use of the Internet-based treatment program will be associated with more cannabis-free days in comparison to only access to information about cannabis use and its harmful effects.

The secondary hypotheses to be tested are:

1. That the use of the Internet-based treatment program will be associated with a larger decline in cannabis consumption (frequency and quantity) among individuals with regular cannabis use in comparison to only access to information about Cannabis use and its harmful effects.
2. That the use of the Internet-based treatment program will be associated with a larger decline in alcohol consumption, depression and anxiety and increased sense of coherence in comparison to only access to information about Cannabis use and its harmful effects.
3. That the proportion of individuals who seek professional help or talk to their relatives or friends about reducing or stopping cannabis use will be greater among those who use the Internet-based treatment program than among those who only have access to information about cannabis use and its harmful effects.

Recruitment procedure and baseline measures Study participants will be recruited through an advertisement on Cannabishjalpen.se. Interested individuals will answer questions about gender, age, country of birth, educational attainment, employment, marital status, living situation, and cannabis use.

The intervention group Individuals randomized to the intervention group will directly after randomization answer questions about alcohol use, use of drugs other than alcohol and cannabis, depression, anxiety, a sense of context and whether they during the last 12 months has received professional help to reduce or quit their cannabis use or during the same period have raised this issue with their relatives or friends.

Further, they will fill out a survey on Internet-based services for individuals who wish to reduce or quit their cannabis use. The study participants will then be informed that they, within two days, will gain access to an internet based treatment program designed to help them quit their cannabis use and that they through the program will have the opportunity to communicate with a therapist. Within the next two days, they will gain access to the internet-based treatment program, they will have access to it for two months and they will be contacted again after three months to answer questions about their cannabis and alcohol use, as well as about other previously mentioned issues.

The control group Individuals randomized to the control group will undergo exactly the same procedure as the intervention group. The difference is that the control group will be informed that they in about three months will gain access to an internet based treatment program designed to help them quit their cannabis use (i.e. when the data collection for follow-up is completed).

Otherwise, participants in both groups will have the opportunity to use factual information that is available to everyone on Cannabishjalpen.se.

Follow-up procedure Study participants who were randomized to the intervention group will have access to intervention in two months. Three months after recruitment to the study, study participants from both groups will get an automated email invitation to participate in the three-month follow-up. The email will include a personalized link that when clicked on will redirect the participant to follow-up page where they will be asked to once again answer questions about their cannabis and alcohol use, depression and anxiety, seeking professional help for cannabis use as well as the help of family or friends and questions about whether they have used any other internet or telephone services to reduce or quit their cannabis use. The entire follow-up procedure will be completed via the internet.

ELIGIBILITY:
Inclusion Criteria:

* Age >15
* Cannabis use 1 time/week or more often during the past six months.

Exclusion Criteria:

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2015-06-26 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Number of days without cannabis use. | Past seven days

SECONDARY OUTCOMES:
Grams of cannabis consumed. | Past three months
Reduction in frequency of cannabis use. | Past three months
Number of DSM-V criteria for cannabis dependence. | Past three months
Total score on Cannabis Abuse Screening Test (CAST). | Past three months
  Total score range 0-24 where higher scores indicate worse outcome.
Receiving professional help for cannabis use from relatives or friends. | Past three months
Receiving help for cannabis use from relatives or friends. | Past three months
Number of standard (alcohol) drinks. | Past seven days.
Total score on Sense of coherence Scale. | Past three months
  Total score range13-91, where higher scores indicate better outcome.
Total score on Montgomery Åsberg Depression Rating Scale - Self reported (MADRS-S). | Past three months
  Total score range 0-60 where higher scores indicate worse outcome.
Total score on Generalized Anxiety Disorder Assessment (GAD-7). | Past three months
  Total score range 0-21 where higher scores indicate worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Sinadinovic, PhD, Principal Investigator — Karolinska Institutet, Department of Clinical Neuroscience, Center for Psychiatric Research and Education
Locations (1):
- Center for Psychiatric Research, Stockholm, Sweden

REFERENCES:
- [Derived] Sinadinovic K, Johansson M, Johansson AS, Lundqvist T, Lindner P, Hermansson U. Guided web-based treatment program for reducing cannabis use: a randomized controlled trial. Addict Sci Clin Pract. 2020 Feb 18;15(1):9. doi: 10.1186/s13722-020-00185-8. PMID 32070417